CLINICAL TRIAL: NCT01586481
Title: Effectiveness and Safety of an Off- Loading Shoe to Improve Healing and Prevention of Recurrence of Neuropathic Diabetic Plantar Foot Ulcers of the Fore Foot: a Prospective Randomised Pilot Study
Brief Title: Off- Loading Shoe to Improve Healing and Prevention of Recurrence of Neuropathic Diabetic Plantar Foot Ulcers
Acronym: SANIBA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: MAYZAUD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P090501
Record Dates: First submitted 2012-04-25; First posted 2012-04-26 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes Mellitus; Diabetic Neuropathic Foot Ulcer
Keywords: Diabetic foot ulcer; Off loading; Compliance; Healing duration; Amputation rate
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- barouk (Active Comparator)
  Interventions: Device: BAROUK
- sanidiab (Experimental)
  Interventions: Device: SANIDIAB

INTERVENTIONS:
Device: SANIDIAB — off-loading shoe
  Arms: sanidiab
Device: BAROUK — old shoe
  Arms: barouk

SUMMARY:
It's a pilot prospective opened multicentric randomised study. We measure the efficiency and the safety of a new concept of off-loading shoe (SANIDIAB) compared with an old one (BAROUK) to treat chronic diabetic foot ulcer which involved a high risks of amputation 64 diabetic patients with a plantar neuropathic ulcer of the fore foot without infection, osteomyelitis or angiopathy, will be included. 32 patients will be treated with SANIDIAB shoe and 32 with BAROUK shoe

DETAILED DESCRIPTION:
Name of the study : SANIBA

Objective:

The gold standard to heal diabetic foot ulcers is complete off-loading. To wear continuously off loading shoe is very difficult The bad compliance of the patients can lead to infection of the ulcer and amputation of the foot.

The purpose of this study is to compare the efficacy of a new concept of off-loading shoe (a pair of SANIDIAB shoes) with a single BAROUK shoe to treat chronic plantar diabetic foot ulcer of the fore foot. The hypothesis is that the new concept is more efficient because of a good off-loading associated with a best compliance to wear the new concept of shoes.

The study will last 18 months with a duration of study of 6 months per patient It's a pilot prospective multicenter randomised study of 64 diabetic patients with a plantar neuropathic ulcer of the fore foot, treated after randomisation by an off loading shoe BAROUK or a pair of off loading shoes SANIDIAB.

Patients will be followed in a diabetic foot department every 14 days until healing and after healing until 6 months after inclusion in the study.

The main outcome measure is the healing duration of the diabetic foot ulcers in both group of treatment.

The secondary outcome measure is the rate of reulceration after healing , the rate of amputation and compliance of patients 64 patients will be included in 2 groups: 32 will wear SANIDIAB shoes and 32 BAROUK shoe.

ELIGIBILITY:
Inclusion criteria :

* More of 18 years old man or woman
* Type 1 or 2 Diabetes mellitus
* A new plantar ulcer of the fore foot or the toes
* GRADE 1A or 2 A of the University of Texas Classification
* Neuropathy assessed by absence of sensation in 10g monofilament test

Exclusion criteria

* Severe angiopathy (Grade 3 of the PEDIS classification)
* Osteomyelitis or cellulitis of the foot
* Transmetatarsal amputation
* Other study in course
* Immunosuppressive drugs, antibiotic therapy,
* Hepatic insufficiency
* No possibility to follow the patients every 14 days
* No state health insurance
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Healing duration of the diabetic foot ulcer | 6 months

SECONDARY OUTCOMES:
Rate of reulceration | 6 months
Rate of amputation | 6 months
Compliance of patients to footwear | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Georges HA VAN, MD, Principal Investigator — APHP
Locations (1):
- Groupe hospitalier Pitié-Salpêtrière, Paris, France